CLINICAL TRIAL: NCT04706884
Title: EFFECT OF CEREBRAL OXYGEN SATURATION ON THE ETIOLOGY OF EARLY POSTOPERATIVE HYPERLACTATEMIA: NEW INDICATION FOR KNOWN MONITORING IN CARDIOPULMONARY BYPASS SURGERY
Brief Title: NEW MONITORING IN DIFFERENTIAL DIAGNOSIS OF HYPERLACTATHEMIA IN CARDIOPULMONARY BYPASS SURGERY
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Sevket Gorgulu, Head of Anesthesiology, Acibadem University
Other Study IDs: ATADEK 2018-2/21
Record Dates: First submitted 2021-01-06; First posted 2021-01-13 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Etiology of Hyperlactathemia; Early Period After Cardiopulmonary Bypass Surgery; Washout Phenomenon
Keywords: Early Hyperlactatemia; Cerebral Oxygen Saturation,; Cardiovascular Surgery
MeSH Terms: conditions — Hyperlactatemia | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Near infrared spectroscopy — The rSO2 (cerebral oxygen satutation) was continuously monitored by NIRS (Near infrared spectroscopy) with a sensor positioned on the forehead of the patient

SUMMARY:
Objective: The objective of the study was to investigate a reverse correlation between blood lactate levels and rSO2, and distinguish between hypoxic and non-hypoxic hyperlactatemia seen in the early postoperative period.

DETAILED DESCRIPTION:
The objective of the prospective study was to investigate a reverse correlation between blood lactate levels and rSO2, and distinguish between hypoxic and non-hypoxic hyperlactatemia seen in the early postoperative period.

Sixty American Society of Anesthesiologists (ASA) II-III patients were included in this study. Perioperative data, including age, weight, body surface area, gender, body temperature, preoperative co-morbidities, intraoperative and postoperative hemodynamic parameters, arterial blood gas analysis (ABG), cardiopulmonary bypass and aortic cross-clamp duration, flow rate, urine output, and blood product and inotropic agent usage, were recorded. Postoperative plasma lactate levels were measured simultaneously with cerebral tissue oxygen saturation (rSO2) in both cerebral hemispheres at 10 different time points.

ELIGIBILITY:
Inclusion Criteria:

* ASA) II-III patients, aged 43-80 years, undergoing on-pump coronary artery bypass grafting

Exclusion Criteria:

* Active congestive cardiac failure, intraoperative death, urgent cardiac surgery or reoperation, hemodynamic instability or need of inotropic support before the operation, the elevation of any parameters preoperatively suggestive of systemic hypoperfusion, coagulopathy, renal failure, hepatic dysfunction, local or systemic infection, and inflammation.

Ages: 43 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo elective bypass surgery and extracorporeal circulation
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Differantial Diagnosis of early hyperlectathemia | through study completion, an average of 1 year
  To understand whether early hyperlactathemia after cardiopulmonary bypass surgery is due to hypoxic or non-hypoxic causes, we will look at the correlation between blood lactate level and cerebral oxygen saturation (rSO2)

CONTACTS AND LOCATIONS:
Overall Officials: Fevzi Toraman, Prof, Study Chair — Acıbadem University School of Medicine Head of Department of Anesthesiology and Reanimation
Locations (2):
- Turkey (Türkiye) (2):
  - Acıbadem Mehmet Ali Aydinlar University Atakent Hospital, Istanbul, Atakent
  - Acibadem University, Istanbul

IPD SHARING:
Plan to Share IPD: No